CLINICAL TRIAL: NCT00910416
Title: The Comparability of Bispectral Index and Neurosense During Total Intravenous Anesthesia and Balanced Anesthesia
Brief Title: The Comparability of Bispectral Index and Neurosense During Anesthesia
Status: Terminated | Type: Observational
Why Stopped: Differences between BIS and Neurosense are important. This study can be terminated.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/22
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
Keywords: Anesthesia; Monitoring, Intraoperative; Electroencephalography/*drug effects
MeSH Terms: interventions — Propofol; Remifentanil; Atracurium; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients receiving iv anesthesia
  Interventions: Drug: propofol, remifentanil, atracurium; Device: EEG monitoring
- patients receiving balanced anesthesia
  Interventions: Drug: propofol, remifentanil, atracurium, sevoflurane; Device: EEG monitoring

INTERVENTIONS:
Drug: propofol, remifentanil, atracurium — propofol, remifentanil, atracurium dosages are adapted according to clinician's judgment
  Groups: patients receiving iv anesthesia
Drug: propofol, remifentanil, atracurium, sevoflurane — dosages are adapted according to clinician's judgment
  Groups: patients receiving balanced anesthesia
Device: EEG monitoring — simultaneous monitoring with Bis and Neurosense

SUMMARY:
The assessment of anesthesia depth was based, until recently, on the evolution of hemodynamic parameters. Nowadays it can be evaluated by several monitoring methods, derived from electroencephalogram analysis, namely the Bispectral Index (Aspect Medical Systems, Newton, USA). A new modality is currently under development: the NeuroSENSE (Cleveland Medical Devices Inc., Cleveland, OH 44103, USA). The goal of this study is to compare both monitoring modalities during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring either intravenous anesthesia or balanced anesthesia (including sevoflurane)

Exclusion Criteria:

* Pregnant women,
* Allergy to propofol, remifentanil, morphine, muscle relaxant, or to a component,
* Hypersensibility to sufentanil, remifentanil or to a derivate of fentanyl,
* History of neurological disorder or central brain lesion, of muscle disease,
* Patient carrying a pacemaker,
* Patients receiving a psychotropic treatment or a morphine agonist-antagonist,
* Alcoholic patients and patients taking opiates,
* Surgery with extracorporeal circulation,
* Surgical position incompatible with an adequate positioning of the probe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Concordance between pairs of Bispectral Index and Neurosense indices during maintenance of anesthesia | at the end of each case
  Statistical analysis of concordance

SECONDARY OUTCOMES:
Concordance between pairs of Bispectral Index and Neurosense indices during induction and emergence | at the end of each case
  Statistical analysis of concordance

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Dept of Anesthesia, Hôpital Foch, Suresnes, France

REFERENCES:
- [Background] Zikov T, Bibian S, Dumont GA, Huzmezan M, Ries CR. Quantifying cortical activity during general anesthesia using wavelet analysis. IEEE Trans Biomed Eng. 2006 Apr;53(4):617-32. doi: 10.1109/TBME.2006.870255. PMID 16602568